CLINICAL TRIAL: NCT02633345
Title: Effects on Tablets Containing Probiotic Candidate Strains on Clinical and Cytokine Markers of Gingival Inflammation and Composition of the Salivary Microbiome
Brief Title: Effects on Tablets Containing Probiotic Candidate Strains
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Mette Kirstine Keller, Assistant Professor, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: H-8-2014-014
Record Dates: First submitted 2015-12-10; First posted 2015-12-17 (Estimated); Last update posted 2016-06-15 (Estimated); Status verified 2016-06

CONDITIONS: Gingivitis
MeSH Terms: conditions — Gingivitis | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Probiotic (Experimental): The probiotic tablets contain Lactobacillus rhamnosus PB01 and Lactobacillus curvatus P2-2 at a dose of 1 * 109 CFU/tablet. The participants will take two tablets a day for four weeks.
  Interventions: Dietary Supplement: Probiotic tablets
- Control (Placebo Comparator): Placebo tablets. The participants will take two tablets a day for four weeks.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic tablets — Tablets with both Lactobacillus rhamnosus PB01 and Lactobacillus curvatus P2-2. Two tablets a day for four weeks
  Arms: Probiotic
Dietary Supplement: Placebo — Placebo tablets
  Arms: Control

SUMMARY:
The aim of the study is to investigate the effect of tablets containing probiotic candidate strains, on gingival inflammation and the levels of selected pro- and anti-inflammatory cytokines in gingival crevicular fluid (GCF). A secondary aim is to describe the effect of the tablets on the salivary microbiome. The null hypothesis is that the clinical measurements, levels of cytokines and microbial composition of saliva will not differ from baseline or between the study and control group.

The study is planned as a double-blind; placebo controlled randomized trial with two parallel arms. The intervention period is planned to be 4 weeks.

80 participants are planned to be enrolled after informed consent and then randomly allocated to either the probiotic group or the placebo group.

The participants are randomly assigned to one of the study groups and given supply of either probiotic tablets or placebo tablets.

The probiotic tablets contain Lactobacillus rhamnosus PB01 and Lactobacillus curvatus P2-2 at a dose of 1 * 109 CFU(Colony Forming Units)/tablet. The participants will take two tablets a day for four weeks. Follow up registrations are conducted after two weeks, four weeks and six weeks.

At each visit, saliva and GCF will be collected and then plaque index (PI)) and bleeding on probing (BOP) will be registered.

All data will be processed with SPSS software (v 22.0; Chicago, Ill, USA). The follow-up values are compared to baseline within each group by Wilcoxon paired two-sided test and differences between groups are analyzed by Wilcoxon unpaired test. A p-value < 0.05 is considered statistical significant.

The participants are fully covered by the patient insurance of The School of Dentistry which cover any damage to the trial participant during the study .There is no expected side effects to the treatment with probiotics. Probiotics are generally considered safe (GRAS: Generally Recognized As Safe) by The European Food Safety Authority (EFSA).

The participants will not benefit directly from the treatment, but the knowledge gained from the study might contribute to the prevention of microbial derived illnesses in the mouth, e.g. caries and periodontitis, in the future. The sample collection does not cause any discomfort to the participants and the tablets have no known side effects. Therefore, the personal benefit of the participants corresponds to the minimal risk and discomfort to the participants.

DETAILED DESCRIPTION:
Background:

The human saliva offers an easy accessible and non-invasive opportunity to study bacterial interactions as well as biomarkers of health and disease. The Human Microbiome Project has provided insights that the biofilms inside and outside our bodies have co-evolved with mankind and play an important role for health. This is also true for the oral cavity in which the microbiota does not play a passive role but actively contributes to the maintenance of oral health. However, certain ecological shifts in the microbiome allow pathogens to manifest and cause oral diseases. According to the ecological plaque hypothesis, caries and periodontitis are the result of environmentally induced overgrowth of aciduric and proteolytic species, respectively.

Bacteriotherapy is the term used when a harmless effector strain is implanted in the host's microflora to maintain or restore a natural microbiome by interference and/or inhibition of other microorganisms, and especially pathogens. This might open up alternative ways of fighting infectious diseases with less harmful side effects and may also help in the treatment of disorders that seem to have nothing to do with bacteria, such as asthma, obesity and diabetes. Probiotic bacteria, defined as "Live microorganisms which, when administered in adequate amounts, confer a health benefit on the host" (WHO), are commonly suggested candidates for bacteriotherapy. The potential mechanisms of action are still not fully understood but it seems clear that there are local (direct) as well as systemic (indirect) effects. According to Reid the potential avenues are: i) co-aggregation with pathogens and growth inhibition, ii) bacteriocin and hydrogen peroxide production, iii) competitive exclusion through antagonistic activities on adhesion sites and nutrition, iv) systemic immunomodulation.

In vitro studies have shown effect on co-aggregation and growth inhibition and clinical studies have shown effect on clinical parameters of gingival inflammation but still little is known about the immunomodulatory effect and the host-microbe interaction.

Periodontal diseases are among the most widespread infectious diseases in man and can lead to tooth loss. If left untreated gingivitis can lead to periodontitis.

The different surfaces of the oral cavity are all continuously bathed in saliva and several pathogenic species in saliva have been associated with periodontal disease. Studies on the microbial effect of probiotic bacteria on oral health have so far been based on conventional cultivation methods and have been focused on one or a few strains. The new high-throughput techniques provide a possibility for more comprehensive and precise picture of the bacterial profiles, but to date only a few studies have used sequencing to determine the bacterial composition of saliva after intake of probiotic bacteria. Most analyze the composition after a very short term intake of the probiotic bacteria. Hence, there is only one study which have analyzed the composition after longer intervention period and correlated this to clinical outcomes.

Aim:

The aim of the study is to investigate the effect of tablets containing probiotic candidate strains, on gingival inflammation and the levels of selected pro- and anti-inflammatory cytokines in gingival crevicular fluid (GCF). A secondary aim is to describe the effect of the tablets on the salivary microbiome. The null hypothesis is that the clinical measurements, levels of cytokines and microbial composition of saliva will not differ from baseline or between the study and control group.

Study design:

The study is planned as a double-blind; placebo controlled randomized trial with two parallel arms. The intervention period is planned to be 4 weeks. The study plan will be submitted for ethical approval.

Material:

The participants will be recruited among patients at the clinic at School of Dentistry and through www.forsogsperson.dk. 80 participants are planned to be enrolled after informed consent and then randomly allocated to either the probiotic group or the placebo group. Sample size was determined by a power analysis (α= 0.05 and β=0.2) based on values of BOP obtained previously. Seventy-four participants are needed and 80 are enrolled in order to compensate for expected drop-outs.

Recruitment: If the participants after reading the notice about the study express interest in the study they will be invited to an information appointment with assistant professor and dentist Mette Kirstine Keller. Prior to the appointment, the participants will be informed that they have the right to bring a companion to the information meeting. They will also receive the written information about the study. The appointment will take place in a meeting room without other people present than the investigator, the participant and possibly a companion. The oral information will be based on the written information and will be given in a plain language without any value-laden terms. The investigator is responsible for ensuring that the participant has understood all given information before the project begins. All comments from the participant are taken into relevant consideration both during the information interview and the study. At any time the participant can withdraw from the project. The informed consent for participation in the trial is given on the basis of oral and written information, and such consent may be given after at least 24 hours of reflection time. The project does not include subjects who, because of physical or mental handicap, cannot give the informed consent.

Methods:

Intervention:

After informed consent, baseline examination and sampling, the participants are randomly assigned to one of the study groups and given supply of either probiotic tablets or placebo tablets.

The probiotic tablets contain Lactobacillus rhamnosus PB01 and Lactobacillus curvatus P2-2 at a dose of 1 * 109 CFU/tablet. The strains are chosen based on in vitro assays investigating growth inhibition of pathogens and immunomodulation. The placebo tablets are identical in size and composition but without the addition of the probiotic strains. Both tablets are provided by Bifodan A/S. The participants will be instructed to take one tablet in the morning and one in the evening thirty minutes after tooth brushing. The tablets are packed in identical pots with color coding. The code will be kept from the investigators until the analysis are finished.

The participants will take two tablets a day for four weeks. Follow up registrations are conducted after two weeks, four weeks and six weeks.

Clinical procedures:

At each visit, saliva and GCF (Gingival Crevicular Fluid) will be collected and then plaque index (PI)) and bleeding on probing (BOP) will be registered. For the collection of GCF, two contralateral buccal sites from the upper incisors, canines or premolars will be selected from each participant. Visual supragingival plaque on the selected teeth will be removed and the sites will be dried with cotton pellets. GCF will be collected using periopaper strips (ProFlow, Amityville, NY, USA) gently inserted in the gingival sulcus for 20 s. The position of the strip is marked on a chart to secure the identical sample site at the follow ups. In case of blood contamination, the strip is discharged and the sampling is repeated after 5 min. The volume of GCF is recorded using a Peritron 8000 (Proflow) and expressed in μL. One strip holds approximately 0.1-0.4 μL GCF. The strips are then transferred to plastic tubes and stored at -80ºC until further analysis.

For the saliva samples, paraffin-stimulated whole saliva is collected during a 3-minute period at least two hours after any food intake. The approximate amount of saliva at normal rate will be 3-6 ml after 3 minutes. The collected saliva is immediately frozen in 1.5 ml aliquots and stored at -80ºC until further analysis. The remainder of the sample will be destroyed after completion of the study.

Laboratory procedures:

Analysis of cytokines on GCF: The absorbed GCF is eluated in 120 μL PBS (phosphate buffered saline) containing 0.05 % Tween 20. The levels of INFγ, TNF-α, IL-8, IL-10 and IL-12 is determined using luminex and multiplex immunoassay panels (LINCOplex, LINCO Research, Inc, USA) in accordance with the manufacturer's manual. The concentrations of the cytokines are expressed as pg/ml.

Analysis of the salivary microbiome: Total bacterial DNA will be extracted from 2 ml of thawed saliva sample for identification and comparison of the composition and stability of the total microbial communities in the two trial groups through amplicon sequencing of the phylogenetic marker gene 16S rRNA. The hypervariable region V3-V4 of bacterial and archaeal 16S rRNA genes will be PCR amplified using specific primers 341F and 806R and analyzed by an established high-throughput sequencing pipeline developed by the University of Copenhagen Microbiology partner based on state-of-the-art sequencing technologies (Illumina Mi-Seq) and custom made bioinformatic tools specifically designed for analysis of large microbiome datasets.

Statistical methods:

All data will be processed with SPSS software (v 22.0; Chicago, Ill, USA). The follow-up values are compared to baseline within each group by Wilcoxon paired two-sided test and differences between groups are analyzed by Wilcoxon unpaired test. A p-value < 0.05 is considered statistical significant.

Data management:

All collected data will be treated in compliance with the Act on Processing of Personal Data and "The Health Law". At inclusion the participants will be assigned a unique number and a separate protocol without personal identification number.

Scientific importance:

The study may provide evidence that the probiotic tablets can influence clinical markers of gingival inflammation and/or pro- and anti-inflammatory cytokines, which can lead to new strategies in managing gingivitis and maintaining oral health. The use of probiotic bacteria in treatment of dental diseases could be one option the use of antibiotics. Furthermore it will provide new insights to the effect of introducing new strains to the salivary microbiome which is supposed to be a significant event in bacteriotherapy.

Risks and Adverse Effects:

The participants are fully covered by the patient insurance of The School of Dentistry which cover any damage to the trial participant during the study .There is no expected side effects to the treatment with probiotics. Probiotics are generally considered safe (GRAS: Generally Recognized As Safe) by The European Food Safety Authority (EFSA).

The participants will be asked to report any unexpected adverse effect.

Ethical considerations:

The participants will not benefit directly from the treatment, but the knowledge gained from the study might contribute to the prevention of microbial derived illnesses in the mouth, e.g. caries and periodontitis, in the future. The sample collection does not cause any discomfort to the participants and the tablets have no known side effects. Therefore, the personal benefit of the participants corresponds to the minimal risk and discomfort to the participants. The participants who complete the trial will be compensated with a gift voucher of 500 DKK to Magasin. It should be emphasized that positive, negative and inconclusive results will be published.

Time Schedule:

Preparation of the study will be carried out in the winter 2014/2015. After ethical approval, patients can be recruited to the study during winter/spring 2015.

ELIGIBILITY:
Inclusion Criteria:

* presence of at least two buccal marginal sites with moderate gingival inflammation according to the Löe index with a probing depth of ≤ 5 mm

Exclusion Criteria:

* regular intake of probiotic bacteria
* smoking
* pregnancy
* intake of antibiotics within the last two months before baseline
* low stimulated saliva rate (0,8 ml/min)
* rampant decay with several untreated caries lesions

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2015-09; Primary Completion 2016-04 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Cytokines in GCF: INFγ, TNF-α, IL-8, IL-10 and IL-12 (ng/uL) | Baseline, two weeks, four weeks, 6 weeks
  Change between timepoints
Plaque Index | Baseline, two weeks, four weeks, 6 weeks
  Change between timepoints. Amount of plaque according to Loe Index
Number of sites with Bleeding on Probing | Baseline, two weeks, four weeks, 6 weeks
  Change between timepoints

SECONDARY OUTCOMES:
Salivary microbiome (ng/UL) | Baseline, two weeks, four weeks, 6 weeks
  Concentration of 200 selected bacteria in saliva. Change between timepoints

CONTACTS AND LOCATIONS:
Locations (1):
- University of Copenhagen, Copenhagen, Denmark